CLINICAL TRIAL: NCT01565057
Title: A Study on the Effect of Gastric Layering and Emptying Induced by a Food Emulsion
Brief Title: Gastric Layering Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Alan Mackie, Principle Investigator, Quadram Institute Bioscience
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IFR07/2010
Record Dates: First submitted 2012-03-23; First posted 2012-03-28 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: emulsion; emptying; protein; layering

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sedimenting meal (Experimental): To assess whether rates of gastric emptying of a specifically formulated emulsion drink are significantly different from a control drink and that this in turn leads to differences in satiation (cessation in the desire to eat) and satiety (desire to limit further food intake) as measured by visual analogue scale (VAS) satiety questionnaire and blood CCK.
  Interventions: Other: sedimenting meal

INTERVENTIONS:
Other: sedimenting meal — The active system quickly forms a sedimenting layer of small particles that contain most of the caloric content of the system. This system is made by adding finely grated cheese (particle size 0.5-2 mm) to yoghurt and consumption is followed by drinking 327 ml water.

SUMMARY:
This comparative study is designed to compare the gastric layering and rates of emptying and by inference rates of digestion of two food emulsions. Two types of dairy based foods will be used, one which will sediment in the stomach and one that will not. On each of two study days, a total of 9 post drink MRI scans will be taken to assess gastric layering and emptying. Cannulation will allow blood samples to be taken periodically for subsequent analysis for the presence of specific digestion related hormones. A total volume of 36 ml of blood will be removed and volunteers will also be asked to complete a questionnaire at predetermined times to assess feelings of satiation.

ELIGIBILITY:
Inclusion Criteria:

* Male (hormonal status of women would introduce more variation within small group)
* Age 20-50y
* BMI 19-30
* Apparently healthy
* Normally eat lunch
* Willing to eat the finely grated cheese meal
* Provide written informed consent

Exclusion Criteria:

* Individuals with an intolerance or allergy to any of the constituents of the test meal
* Smokers or smoked within the last year (smoking affects satiety/hunger)
* Diagnosed with any long term illness requiring active treatment e.g. diabetes, cancer, cardiovascular disease
* Have had surgery on the stomach or intestine or suffered from gastrointestinal disease, whether diagnosed or self reported
* Regular (more than once in 10 days) use of antacids, laxatives
* Any problems with swallowing
* Take prescription medication for digestive or gastrointestinal conditions.
* Volunteers taking part in another study (other than a questionnaire based study).
* Blood pressure greater than 160/100 or less than 90/50 or 95/55 if symptomatic.
* Individuals with special dietary requirements (eg vegetarians)
* If attended a study during the previous four months where combined blood sampling from previous study and present study would exceed 470mL.
* If any of the clinical screening results are indicative of a health problem which would affect the volunteers well-being or which would affect the study data.
* Refusal to give permission to inform GP of participation in study
* Recent unexplained weight gain or loss
* History of back problems or any other condition which limit ability to repeatedly sit up and lie down
* Hiatus Hernia
* MRI scanning specific exclusion criteria

  * Cardiac pacemaker or artificial heart valve
  * Any surgery in the last 6 months
  * Aneurysm clips (metal clips from surgery)
  * Implant, pump or any medical device in the body (eg cochlear implant, neurostimulator, intra-venticular shunt)
  * Worked with metals (using lathes or grinders) or sustained injury to eyes involving metal splinters or fillings
  * Have artificial eyes or limbs
  * Have been injured with shrapnel or bullets
  * Suffer from fits, blackouts or epilepsy
  * Claustrophobia sufferer

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rates | 3 hours
  The primary objective is to measure gastric emptying rates and layering patterns as a function of time in healthy volunteers using two different meals, one which sediments gastric digestion and one in which it does not.

SECONDARY OUTCOMES:
Fullness and satiety from visual analogue scores | 3.5 hours
  To correlate gastric emptying rates with satiety responses after the meal
levels of CCK in the blood | 3.5 hours
  To correlate gastric emptying rates with levels of the GI hormone CCK in blood

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Mackie, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom